CLINICAL TRIAL: NCT04015362
Title: Pulsed Magnetic Stimulation - Managing Spasticity in Spinal Cord Injury
Acronym: OsStim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RL1 535
Record Dates: First submitted 2019-04-26; First posted 2019-07-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed magnetic stimulation of the spinal cord (Experimental): Sub-threshold intermittent pulsed magnetic stimulation of spinal cord
  Interventions: Procedure: Sub-threshold intermittent pulsed magnetic stimulation
- Sham magnetic stimulation (Sham Comparator): Sham - patient and machinery placed in same position as intervention arm but no magnetic stimulation delivered
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Sub-threshold intermittent pulsed magnetic stimulation — Application of sub-threshold intermittent pulsed magnetic stimulation to spinal cord
  Arms: Pulsed magnetic stimulation of the spinal cord
Procedure: Sham — Application of sham magnetic stimulation to spinal cord
  Arms: Sham magnetic stimulation

SUMMARY:
Spasticity (tightening, spasming and/or contractions of muscles) is a commonly encountered consequence of injuries to the central nervous system. Spasticity has an adverse effect on quality of life and function of patients with spinal cord injuries, stroke and cerebral palsy. Conventional management consists of medication, injections of botulinum toxin and occasionally extensive surgical interventions. Several studies have examined the use of repetitive magnetic stimulation of the brain and of peripheral nerves to produce long-term depression of spasticity. Recently, Theta burst sequence low-dose magnetic stimulation has been shown to mark unused synaptic connections for deletion. By using pulsed magnetic stimulation of the spinal cord the abnormal connections arising from injury may be identified for deletion, therefore potentially minimising the mis-firing circuits.

The investigators plan, in this pilot study, to test whether firstly the application of pulsed magnetic stimulation of the spinal cord is achievable in patients with spinal cord injury (SCI) and secondly whether it has an effect on lower limb spasticity.

These results will be used to help design a larger trial, to expand the numbers of participants and variety of pathologies treated.

Participants (in-patients at the Midland Centre for Spinal Injuries) with stable SCI will be randomised to receive either intermittent pulsed magnetic stimulation or no stimulation. Patients will be blinded as to whether they are receiving stimulation (the machine will be active up and placed in the same position for both groups, except the sham group will have the stimulation coil applied in an orientation that does not deliver the magnetic field to the spinal cord).

DETAILED DESCRIPTION:
The investigators are trying to understand the potential for low-dose magnetic stimulation to reduce unwanted symptoms including spasticity following a spinal cord injury. After an injury to the spinal cord the nerves within the spinal cord below the level of the injury reorganise themselves. This leads to unwanted connections producing a condition known as spasticity. Spasticity is experienced by patients as unwanted muscle stiffness. In patients with some sensation this can cause pain and can often lead to problems with bones and joints and difficulties with positioning for seating and standing. Along with spasticity, altered functioning in the nerves that control blood pressure, sweating, bowel and bladder can all create difficulties for someone who has had such an injury.

It is now known that the nervous system reorganises itself on a continuous basis even after humans have finished growing. For example, it has to do this so that we can form memories and learn. This process is necessary in healthy life and is regulated by an army of cells that roam through the central nervous system including the spinal cord. These cells known as microglial cells act as gardeners, pruning connections that aren't needed and strengthening connections that are needed. From recent work in the field of biology it is now understood that a chemical called complement is used as a marker a bit like paint on a tree that is to be trimmed, to tell the microglial cells where to cut or where to strengthen. Very low level pulsed magnetic stimulation can mark connections that need to be trimmed so that the microglial cells can go about their job. The investigators want to identify whether by using a very low dose of magnetic stimulation we could reduce the abnormal connections in the spinal cord that cause spasticity. The investigators believe this is a very safe treatment because it is using magnetic stimulation on the spinal cord at a 10th of the level that is commonly used on the brain.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Aged above 18 years and below 99 years old
* Possesses mental capacity
* Established spinal cord injury Frankel grade A, B or C, at least 2 months prior to recruitment
* Involvement of the spinal cord at L1 level or above
* Admitted to the Midland Centre for Spinal Injuries (Oswestry, UK)
* Expected to remain an in-patient for the duration of the study
* Experiences spasticity affecting the lower limbs

Exclusion Criteria:

* Pregnant
* Non-MRI compatible spinal fixation in place
* Implanted Insulin pump
* Change of spasticity medication within last 2 weeks
* Planned spasticity intervention at this admission
* Epilepsy with fit within the last 12 months
* Currently taking donezipil hydrochloride
* Currently taking sodium valproate
* Cardiac Pacemaker or wires
* Internal cardioverter defibrillator (ICD)
* Deep Brain Stimulator
* Tattoo on lower back
* Radioactive seeds
* Cochlear implant/ear implant
* Vagus nerve stimulator (VNS)
* Intrathecal Baclofen Pump
* presence of shrapnel, bullets, pellets, Ball bearings in the patient's body
* Wearable cardioverter defibrillator
* Surgical clips, staples or sutures
* VeriChip microtransponder
* Wearable infusion pump
* Irremovable Body piercings

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Modified Penn Spasticity scale | Baseline (up to 24 hours before treatment)
  A two-part patient self-reported measure assessing frequency and severity of muscle spasms. Part one asks the patient to describe the intensity and frequency of muscle spasms in the previous 24 hours and part two asks the patient to describe the intensity and frequency of muscle spasms in the previous 1 hour. Frequency is assessed on a 5 point scale ranging from no spasms (0) to spontaneous spasms occurring more than 10 times in the hour (5). Intensity it marked on a 3 point scale of mild, moderate and severe. The higher the scores, the more frequent and the more severe the spasms.
Modified Penn Spasticity scale | Day 14 post start of treatment
  A two-part patient self-reported measure assessing frequency and severity of muscle spasms. Part one asks the patient to describe the intensity and frequency of muscle spasms in the previous 24 hours and part two asks the patient to describe the intensity and frequency of muscle spasms in the previous 1 hour. Frequency is assessed on a 5 point scale ranging from no spasms (0) to spontaneous spasms occurring more than 10 times in the hour (5). Intensity it marked on a 3 point scale of mild, moderate and severe. The higher the scores, the more frequent and the more severe the spasms.
Modified Penn Spasticity scale | Day 28 post start of treatment
  A two-part patient self-reported measure assessing frequency and severity of muscle spasms. Part one asks the patient to describe the intensity and frequency of muscle spasms in the previous 24 hours and part two asks the patient to describe the intensity and frequency of muscle spasms in the previous 1 hour. Frequency is assessed on a 5 point scale ranging from no spasms (0) to spontaneous spasms occurring more than 10 times in the hour (5). Intensity it marked on a 3 point scale of mild, moderate and severe. The higher the scores, the more frequent and the more severe the spasms.

SECONDARY OUTCOMES:
Pain score | Baseline (up to 24 hours before treatment)
  A patient self-reported score of pain, as published in the Spinal Cord journal 2008 (46:818-823).
  Patients are initially asked whether they have had any pain in the last 7 days, including today. If no, then no further questions are asked. If yes, they are asked how many different pain problems they had (1, 2, 3, 4 or >5) and then to subsequently describe their 3 worst pain problems. Location, intensity and length of pain are then recorded. Further, questions with a scale of 0 (not at all) to 6 (extreme interference) are asked about how the patients' pain affects their daily activities, mood and sleep.
Pain score | Day 14 post start of treatment
  A patient self-reported score of pain, as published in the Spinal Cord journal 2008 (46:818-823).
  Patients are initially asked whether they have had any pain in the last 7 days, including today. If no, then no further questions are asked. If yes, they are asked how many different pain problems they had (1, 2, 3, 4 or >5) and then to subsequently describe their 3 worst pain problems. Location, intensity and length of pain are then recorded. Further, questions with a scale of 0 (not at all) to 6 (extreme interference) are asked about how the patients' pain affects their daily activities, mood and sleep.
Pain score | Day 28 post start of treatment
  A patient self-reported score of pain, as published in the Spinal Cord journal 2008 (46:818-823).
  Patients are initially asked whether they have had any pain in the last 7 days, including today. If no, then no further questions are asked. If yes, they are asked how many different pain problems they had (1, 2, 3, 4 or >5) and then to subsequently describe their 3 worst pain problems. Location, intensity and length of pain are then recorded. Further, questions with a scale of 0 (not at all) to 6 (extreme interference) are asked about how the patients' pain affects their daily activities, mood and sleep.
Ashworth score | Baseline (up to 24 hours before treatment)
  A clinician assessed score of muscle tone in the hamstring, quadriceps and triceps surae. Flexion or extension of the joint is tested to score muscle tone throughout the range of motion on a scale of 0 (no increase in muscle tone) to 4 (muscle rigid). The higher the score, the more muscle spasticity is indicated.
Ashworth score | Day 14 post start of treatment
  A clinician assessed score of muscle tone in the hamstring, quadriceps and triceps surae. Flexion or extension of the joint is tested to score muscle tone throughout the range of motion on a scale of 0 (no increase in muscle tone) to 4 (muscle rigid). The higher the score, the more muscle spasticity is indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Roberts, FRCS, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom